CLINICAL TRIAL: NCT04389749
Title: The Role of Continuous Passive Motion in Pain Control of Patients Undergoing Operative Management of Isolated Acetabular Fractures, Supracondylar Femur Fractures, or Tibial Plateau Fracture: a Comparative Study
Brief Title: Continuous Passive Motion Following Fixation of Pelvic and Knee Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, H. Claude Sagi, MD, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OS19088 IRB 2019-0541
Record Dates: First submitted 2020-04-26; First posted 2020-05-15 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Fractures, Bone
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Intervention Model Description: prospective comparative cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CPM (Experimental): The experimental group will have a CPM applied in the PACU immediately post-op and it will be utilized while the patient is awake in bed for 2 hours on and 2 hours off, when not mobilizing with Physical Therapy (PT). The experimental group will also have traditional PT, including sessions 1 to 3 times a week.
  Interventions: Device: CPM
- No CPM (No Intervention): The control group will have typical care, including working with physical therapy 1 to 3 times a week.

INTERVENTIONS:
Device: CPM — CPM-continuous passive motion device.
  Arms: CPM

SUMMARY:
The investigators will directly compare the visual analog scale scores and narcotic pain medication requirements in the patients who have continuous passive motion (CPM) versus those who do not during the course of the hospital admission following an open reduction internal fixation surgery for acetabular fracture, supracondylar femur fracture, or a tibial plateau fracture.

DETAILED DESCRIPTION:
This will be a prospective comparative cohort study analyzing the practices of three surgeons, one of whom routinely uses CPM following fixation of pelvic and acetabular fractures, and two surgeons who do not.

All patients, over the age of 18 years who have undergone open reduction and internal fixation (ORIF) of isolated acetabular fractures, supracondylar femur fractures, or tibial plateau fracture will be asked to participate. Those who consent will be randomized into two groups. The experimental group will have a CPM applied in the PACU immediately post-op and it will be utilized while the patient is awake in bed for 2 hours on and 2 hours off, when not mobilizing with Physical Therapy (PT). The experimental group will also have traditional PT, including sessions 1 to 3 times a week. The control group will have typical care, including working with physical therapy 1 to 3 times a week. The investigators will directly compare the VAS scores and narcotic pain medication requirements in the patients who have CPM versus those who do not during the course of the hospital admission. VAS scores will be assessed throughout the day by RN and/or PT. Functional outcomes will be assessed at the one-year mark using the Iowa and Majeed pelvic functional outcome tools along with the SF-12. Orthopedic Resident or Nurse Clinical will check the patient for incision integrity each day and each session of using the CPM, the patient will be monitored for adverse events. Data will be collected using Epic.

The investigators will record patient demographics including age, sex, and pre-existing narcotic usage. Fracture type according to the Orthopaedic Trauma Association will be recorded. VAS scores and pain medication requirements will be recorded from the first 48 hours during the patient's stay. Pain scores and CPM use will be obtained from Epic using the flowsheet.

Functional outcomes will be assessed at the one-year mark using the Iowa and Majeed pelvic functional outcome tools along with the SF-12.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater
* Isolated acetabular fractures, supracondylar femur fractures, or tibial plateau fracture
* Have undergone operative intervention for fracture

Exclusion Criteria:

* Injury to either lower extremity that affects the patient's ability to weight bear
* Under the age of 18
* Pregnant
* A prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
VAS Pain Score | Visual Analog Score for pain will be recorded daily after the surgery each day until the patient is discharged or up to 365 days..
  Pain will be assessed by the patient on a scale of 1-10 during hospitalization. 1=no pain; 10=worst pain

SECONDARY OUTCOMES:
SF-12 | This score will be completed at the one-year post-operative visit.
  The Short Form 12 (SF-12) uses just 12 questions to measure functional health and well-being from the patient's point of view. An algorithm is used to generate the physical and mental health composite scores for comparison to normative data. The mean score is set to 50. Scores >50 indicate better physical or mental health than to mean. Scores <50 indicate worse physical or mental health than the mean.

CONTACTS AND LOCATIONS:
Overall Officials: Henry C Sagi, MD, Principal Investigator — University of Cincinnati
Locations (1):
- Univrsity of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No